CLINICAL TRIAL: NCT00270933
Title: Marquis/Maximo VR ICD Programming Practices Registry (MAVRIC VR ICD Registry)
Brief Title: MAVRIC VR ICD Registry
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Other Study IDs: 232
Record Dates: First submitted 2005-12-28; First posted 2005-12-29 (Estimated); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Ventricular Tachycardia; Ventricular Fibrillation
Keywords: defibrillators; LLECG; ventricular tachycardia; ventricular fibrillation
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation | interventions — Registries

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Device: Registry

SUMMARY:
The purpose of this registry is to collect information on the health status of patients receiving Marquis/Maximo VR Implantable Cardiac Defibrillators (ICDs), how the devices are being programmed and how this correlates to clinical patient outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Patients implanted with a new or replacement Marquis VR or Maximo VR ICD

Exclusion Criteria:

* Patients enrolled in a device study that affects treatment and/or programming

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 742
Dates: Start 2004-01; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: George Klein, M.D., Principal Investigator — London H.S.C. University Campus
Locations (91):
- United States (81):
  - Birmingham, Alabama
  - Tuscaloosa, Alabama
  - Little Rock, Arkansas
  - Bakersfield, California
  - Banning, California
  - Fresno, California
  - Mission Viejo, California
  - Sacramento, California
  - San Diego, California
  - Stanford, California
  - Littleton, Colorado
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Jacksonville, Florida
  - Lakeland, Florida
  - Miami Beach, Florida
  - Port Charlotte, Florida
  - St. Petersburg, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Decatur, Georgia
  - Chicago, Illinois
  - Hobart, Indiana
  - Indianapolis, Indiana
  - Cedar Rapids, Iowa
  - Davenport, Iowa
  - Kansas City, Kansas
  - Lexington, Kentucky
  - Owensboro, Kentucky
  - Marrero, Louisiana
  - Baltimore, Maryland
  - Salisbury, Maryland
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Saint Joseph, Michigan
  - Southfield, Michigan
  - Coon Rapids, Minnesota
  - Saint Cloud, Minnesota
  - Jackson, Mississippi
  - Cape Girardeau, Missouri
  - Joplin, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Missoula, Montana
  - Las Vegas, Nevada
  - Lebanon, New Hampshire
  - Englewood, New Jersey
  - Albany, New York
  - Huntington, New York
  - New Hyde Park, New York
  - New York, New York
  - Syracuse, New York
  - Pinehurst, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Mayfield Hts, Ohio
  - Youngstown, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Eugene, Oregon
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Spartanburg, South Carolina
  - Chattanooga, Tennessee
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Corpus Christi, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Odessa, Texas
  - Tyler, Texas
  - Charlottesville, Virginia
  - Richmond, Virginia
  - Tacoma, Washington
  - Milwaukee, Wisconsin
- Canada (10):
  - Edmonton, Alberta
  - Victoria, British Columbia
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Kingston, Ontario
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Ste-Foy, Quebec